CLINICAL TRIAL: NCT02873676
Title: Prevalence and the Effect of Lifestyle Modification Project (LMP) on Clinical Outcomes and Cost-effectiveness Ratio for Sarcopenia in Chinese Adults and Elderly: a Multicenter Randomized Controlled Trail
Brief Title: Prevalence and Effect of Lifestyle Modification on Clinical Outcomes and Cost-effectiveness Ratio for Sarcopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PUMCH344801
Record Dates: First submitted 2015-09-16; First posted 2016-08-19 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Sarcopenia
Keywords: prevalence; lifestyle modification; clinical outcomes
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- nutritional intervention (Experimental): This group received multi-dimensional intensive nutritional intervention for 3 month, which included whey (30g/d,plus three times every week ),vitamin D (1000IU) and omega-3 fatty acid (DHA 1200mg and EPA 800mg).
  Interventions: Behavioral: nutritional intervention
- resistance training program (Experimental): This group received resistance training program which is made up warm-up exercise, muscle strength training and relaxing.
  Interventions: Behavioral: resistance training program
- lifestyle modification project (Experimental): This group receive multi-dimensional intensive nutritional intervention and resistance training program.
  Interventions: Behavioral: lifestyle modification project
- control (Placebo Comparator): This group receive nutritional consulting,which involve dietary pattern modification and protein intake standardization.
  Interventions: Behavioral: control

INTERVENTIONS:
Behavioral: nutritional intervention — The intervention is made up of nutrition supplements and dietary pattern modification, which includes whey 30g/d(plus three times every week),vitamin D 1000IU, omega-3 fatty acid (DHA1200mg and EPA 800mg)
  Arms: nutritional intervention
Behavioral: resistance training program — The training program involve warm-up exercise, muscle strength training and relaxing
  Arms: resistance training program
Behavioral: lifestyle modification project — Lifestyle modification project is made up of multi-dimensional intensive nutritional intervention and resistance training
  Arms: lifestyle modification project
Behavioral: control — The intervention involve dietary pattern modification and protein intake standardization
  Arms: control

SUMMARY:
The purposes of this study were to investigate the prevalence and risk factors for sarcopenia in Chinese adults and elderly, and evaluate the effect of Lifestyle Modification Project (LMP) on Clinical Outcomes, Quality of Life and Cost-effectiveness Ratio.

ELIGIBILITY:
Inclusion Criteria:

* age>=18 year The participants must have basic cognitive function and communication Must be able to provide a written informed consent

Exclusion Criteria:

* age<18 year Concurrent severe cardiac disease, unstable diabetes mellitus,uncontrolled chronic disease,liver and renal failer, which may significantly interfere with study compliance.

Participants received any drugs or supplements known to influence effcet size,such as protein powder, calcium, or vitamin D before the 3 months preceding the study. Participants with electronic or mental device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-03; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
relative skeletal muscle index | 3 months
  RSMI(Unit: kg/m2)is defined as muscle mass

SECONDARY OUTCOMES:
Hand grip | 3 months
  HG(Unit: kg)is defined as muscle strength
gait speed | 3 months
  GP(Unit: s)is defined as physical activity level
quality of life on EQ-5D scale | 3 months
  Scores range from 0 [worse] to 1[best](Unit on a scale)
The rate of fracture | 3 months
  rate of participants with fracture due to fall(Unit: %)
the change of physical function on frail index | 3 months
  Scores range from 0 [normal] to 1[unhealth](Unit on a scale)
the rate of infection complication | 3 months
  Rate of participants with infection complication due to sarcopenia(Unit: %)
mortality rate | 3 months
  Rate of participants mortality(Unit: %)
medical cost on cost-effectiveness ratio | 3 months
  the lower cost，the higher effectiveness(Unit: %)

CONTACTS AND LOCATIONS:
Overall Officials: Kang Yu, Study Chair — Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

REFERENCES:
- [Derived] Li CW, Li Q, Liu Y, Zhang Y, Wang ZK, Xing Y, Niu YS, Pang Y, Yu K. Sarcopenic obesity exacerbates gastric cancer prognosis via increased intermuscular and visceral fat accumulation. Eur J Med Res. 2025 Oct 22;30(1):1012. doi: 10.1186/s40001-025-03251-6. PMID 41126316
- [Derived] Li Z, Cui M, Yu K, Zhang XW, Li CW, Nie XD, Wang F. Effects of nutrition supplementation and physical exercise on muscle mass, muscle strength and fat mass among sarcopenic elderly: a randomized controlled trial. Appl Physiol Nutr Metab. 2021 May;46(5):494-500. doi: 10.1139/apnm-2020-0643. Epub 2020 Nov 20. PMID 33216623
- [Derived] Li CW, Yu K, Shyh-Chang N, Li GX, Jiang LJ, Yu SL, Xu LY, Liu RJ, Guo ZJ, Xie HY, Li RR, Ying J, Li K, Li DJ. Circulating factors associated with sarcopenia during ageing and after intensive lifestyle intervention. J Cachexia Sarcopenia Muscle. 2019 Jun;10(3):586-600. doi: 10.1002/jcsm.12417. Epub 2019 Apr 10. PMID 30969486